CLINICAL TRIAL: NCT02303340
Title: Diagnosis of Decreased Bone Density by Dental Cone Beam Computed Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Ben-Zion Joshua, MD, Otolaryngology Department, Soroka University Medical Center
Other Study IDs: sor 0130-13-ctil
Record Dates: First submitted 2014-11-20; First posted 2014-11-27 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Osteoporosis
Keywords: Cone Beam Computed Tomography; Para Thyroid Hormone; Dual Energy X-ray Absorptiometry; Digital Imaging and Communication in Medicine
MeSH Terms: conditions — Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: Any patient who enrolled and signed informed consent will be sent to bone mineral density DEXA Scan, and for blood testing for PTH, Phosphor, Calcium ,Vitamin D and Creatinine levels. Density measurements will be done in specific sites on the CBCT's of the jaws.
  Interventions: Radiation: Dual Energy X-ray Absorptiometry

INTERVENTIONS:
Radiation: Dual Energy X-ray Absorptiometry
  Other Names: DEXA

SUMMARY:
The purpose of this study is to elucidate the role of Dental Cone Beam Computed Tomography (CBCT) in assessment of bone density. The study population contains men and women above the age of 60 years, eligible for Bone Density Testing in accordance with their health insurance, who underwent a Dental CBCT recommended by their Dental Practitioner. Any patient (eligible for bone density screening by age criteria) undergoing CBCT of either one of the jaws (or both) due to dental reasons, will be sent to a bone mineral density DEXA Scan, and for blood testing for PTH, Phosphor, Calcium ,Vitamin D and Creatinine levels.

Density measurements will be done in specific sites on the CBCT's of the jaws. These measurements will be correlated with the blood tests and DEXA scan results.

DETAILED DESCRIPTION:
The purpose of this study is to elucidate the role of Dental Cone Beam Computed Tomography in assessment of bone density.

The study population contains men and women above the age of 60 years, eligible for Bone Density Testing in accordance with their health insurance, who underwent a Dental CBCT recommended by their Dental Practitioner. Any patient (eligible for bone density screening by age criteria) undergoing CBCT of either one of the jaws (or both) due to dental reasons, will be sent to dual energy x-ray absorptiometry (DEXA) Scan, and for blood testing for parathormone (PTH), Phosphor, Calcium ,Vitamin D and Creatinine levels.

The investigators estimate thousands of Dental Cone Beam Computed Tomographies are being ordered every year, due to dental needs in Israel. In this preliminary prospective pilot study the investigators will evaluate 50 subjects who underwent both Dental CBCT and DEXA scan as a preliminary testing.

Density measurements will be done in specific sites on the CBCT's of the jaws. These measurements will be correlated with the blood tests and DEXA scan results.

The outcomes of this study are:

1. Bone density measurement on Dental CBCT can be used for diagnosis of low bone mass conditions.
2. There is an association between bone density DEXA results, blood tests for Calcium, Phosphor, PTH and Vitamin D and Bone density measurements on Dental CBCTs.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women above the age of 60 years.
2. Underwent Dental Cone Beam Tomography for dental reasons, up to three months before screening.
3. Patients underwent bone density examination at Soroka Medical Center only, during the last year prior commencing the research will be eligible for participation without the need for an additional bone density scanning.

Exclusion Criteria:

1. Patients with current or past treatment of any osteoporotic medication: Alendronate (Alendronate teva, Fosamax, Maxibone , Fosalan, Fosavance), Residronate (Actonel. Ribone), Zoledronic acid (Aclasta, Zomera), Denosumab (Prolia), Teriperatide (Forteo),Raloxifen ( Evista), Stronsium Ranelate (Protelos).
2. Patients taking Corticosteroid Therapy.
3. Patients with history of Head and Neck Neoplasia or Head and Neck Irradiation or Bone Metastasis.
4. Patients with hard tissue pathology of the jaws.
5. Patients after laminectomy and or fixation of lumbar vertebrae or after bilateral hip replacement.
6. Diagnosis of primary hyperparathyroidism.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women above the age of 60 years, eligible for Bone Density Testing in accordance with their health insurance, who underwent a Dental CBCT recommended by their Dental Practitioner.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have Osteoporosis that was shown on the dental CT and the DEXA exams | 12 months

SECONDARY OUTCOMES:
Association between bone density DEXA results, blood tests for Calcium, Phosphor, PTH and Vitamin D and Bone density measurements on Dental CBCTs | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Lindsay R, Cosman F. Chapter 354. Osteoporosis. In: Longo DL, Fauci AS, Kasper DL, Hauser SL, Jameson JL, Loscalzo J, eds. Harrison's Principles of Internal Medicine. 18th ed. New York: McGraw-Hill; 2012.
- [Background] Scarfe WC, Farman AG, Sukovic P. Clinical applications of cone-beam computed tomography in dental practice. J Can Dent Assoc. 2006 Feb;72(1):75-80. PMID 16480609
- [Background] Valiyaparambil JV, Yamany I, Ortiz D, Shafer DM, Pendrys D, Freilich M, Mallya SM. Bone quality evaluation: comparison of cone beam computed tomography and subjective surgical assessment. Int J Oral Maxillofac Implants. 2012 Sep-Oct;27(5):1271-7. PMID 23057044
- [Background] Padbury AD Jr, Tozum TF, Taba M Jr, Ealba EL, West BT, Burney RE, Gauger PG, Giannobile WV, McCauley LK. The impact of primary hyperparathyroidism on the oral cavity. J Clin Endocrinol Metab. 2006 Sep;91(9):3439-45. doi: 10.1210/jc.2005-2282. Epub 2006 Jul 5. PMID 16822829
- [Background] Hastar E, Yilmaz HH, Orhan H. Evaluation of mental index, mandibular cortical index and panoramic mandibular index on dental panoramic radiographs in the elderly. Eur J Dent. 2011 Jan;5(1):60-7. PMID 21228957
- [Background] Neves FS, Oliveira LS, Torres MG, Toralles MB, da Silva MC, Campos MI, Campos PS, Crusoe-Rebello I. Evaluation of panoramic radiomorphometric indices related to low bone density in sickle cell disease. Osteoporos Int. 2012 Jul;23(7):2037-42. doi: 10.1007/s00198-011-1810-z. Epub 2011 Oct 18. PMID 22006042
- [Background] Taguchi A. Triage screening for osteoporosis in dental clinics using panoramic radiographs. Oral Dis. 2010 May;16(4):316-27. doi: 10.1111/j.1601-0825.2009.01615.x. Epub 2009 Aug 7. PMID 19671082
- [Background] Halling A, Persson GR, Berglund J, Johansson O, Renvert S. Comparison between the Klemetti index and heel DXA BMD measurements in the diagnosis of reduced skeletal bone mineral density in the elderly. Osteoporos Int. 2005 Aug;16(8):999-1003. doi: 10.1007/s00198-004-1796-x. Epub 2004 Dec 17. PMID 15605191
- [Background] Mah P, Reeves TE, McDavid WD. Deriving Hounsfield units using grey levels in cone beam computed tomography. Dentomaxillofac Radiol. 2010 Sep;39(6):323-35. doi: 10.1259/dmfr/19603304. PMID 20729181
- [Background] Romme EA, Murchison JT, Phang KF, Jansen FH, Rutten EP, Wouters EF, Smeenk FW, Van Beek EJ, Macnee W. Bone attenuation on routine chest CT correlates with bone mineral density on DXA in patients with COPD. J Bone Miner Res. 2012 Nov;27(11):2338-43. doi: 10.1002/jbmr.1678. PMID 22692725